CLINICAL TRIAL: NCT04587778
Title: Imaging Neural Correlates of Antidepressant Action of Ketamine Stereoisomers Using Pharmacological PET/MR Imaging and Metabolite Analysis.
Brief Title: Imaging Neural Correlates of Ketamine Using PET/MR
Acronym: RSKet
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, Prof., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: v2_06.02.2024
Record Dates: First submitted 2020-09-28; First posted 2020-10-14 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: Ketamine
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine; Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Esketamine ((S)-Ketamine) (Experimental): Single-blind placebo (saline) infusion will be performed during the first PET/MR scan in all subjects, i.e. both arms.
  In a cross-over study design, esketamine will be administered during the second scan and racemic ketamine during the third scan.
  Interventions: Drug: Ketamine Hydrochloride; Drug: Esketamine; Drug: Placebo
- Racemic ketamine ((R,S)-Ketamine) (Experimental): Single-blind placebo (saline) infusion will be performed during the first PET/MR scan in all subjects, i.e. both arms.
  In a cross-over study design, racemic ketamine will be administered during the second scan and esketamine during the third scan.
  Interventions: Drug: Ketamine Hydrochloride; Drug: Esketamine; Drug: Placebo
- Pilot study II: Esketamine ((S)-Ketamine) (Experimental): In a cross-over study design, esketamine will be administered during the first scan and placebo during the second scan.
  Interventions: Drug: Pilot study II: Esketamine; Drug: Pilot study II: Placebo

INTERVENTIONS:
Drug: Ketamine Hydrochloride — intravenous infusion
  Other Names: Racemic ketamine (R, S)-Ketamine
  Arms: Esketamine ((S)-Ketamine); Racemic ketamine ((R,S)-Ketamine)
Drug: Esketamine — intravenous infusion
  Other Names: (S)-Ketamine
  Arms: Esketamine ((S)-Ketamine); Racemic ketamine ((R,S)-Ketamine)
Drug: Placebo — intravenous infusion
  Other Names: saline solution
  Arms: Esketamine ((S)-Ketamine); Racemic ketamine ((R,S)-Ketamine)
Drug: Pilot study II: Esketamine — intravenous infusion
  Other Names: (S)-Ketamine
  Arms: Pilot study II: Esketamine ((S)-Ketamine)
Drug: Pilot study II: Placebo — intravenous infusion
  Other Names: Saline solution
  Arms: Pilot study II: Esketamine ((S)-Ketamine)

SUMMARY:
The purpose of this randomized, placebo-controlled study is to investigate pharmacodynamic differences between racemic ketamine and esketamine using functional fluorodeoxyglucose ([18F]FDG) positron emission tomography/magnetic resonance imaging (PET/MR)

Pilot study I:

A pilot study with healthy controls will be performed in order to investigate pharmacokinetic behavior and acute behavioral effects of intravenous ketamine infusion.

Pilot study II:

A pilot study including 15 healthy volunteers will be performed in order to optimize scanning procedures. The pilot study follows a randomized, placebo-controlled, double-blind, cross-over study design. After enrollment into the study all subjects will undergo two [18F]FDG PET/CT scans in the course of which they will receive either S-ketamine or placebo during the first scan and the respective other study medication during the second scan.

ELIGIBILITY:
Inclusion Criteria:

* General health based on medical history, physical examination and structured clinical interview for the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) (SCID)
* Age 18 to 55 years
* Right-handedness (due to potential lateralization effects of lefthanded subjects)
* Willingness and competence to sign the informed consent form.

Exclusion Criteria:

* Current or history of psychiatric or neurological disease
* Current medical illness requiring treatment
* Pregnancy or current breastfeeding
* Current or former substance abuse
* Diagnosis of an Axis-1 psychotic disorder in a first-degree relative
* Any contraindication for MRI (e.g., MR incompatible implants, etc.) including dental implants causing signal artifacts
* For subjects participating in earlier studies using ionizing radiation, the total radiation exposure of 30 millisievert (mSv) over the last 10 years must not be exceeded, as specified in the Austrian legislation on radiation protection (www.ris.bka.gv.at). Accordingly, body weight >100kg is an exclusion criterion (5.1 Megabequerel (MBq)/kg * 100kg * 0.019 mSv/MBq* 0.885 = 8.58 mSv per scan, the factor 0.885 is considered due to continuous radioligand infusion, see PET scanning).
* Failure to comply with the study protocol or to follow the instruction of the investigating team.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cerebral metabolic rate of glucose (CMRGlu) | during PETMR/during 45 minutes of infusion
  Change in CMRGlu between each PET/MR scan
Change in cerebral blood flow (CBF) | during PETMR/during 45 minutes of infusion
  Change in CMRGlu between each PET/MR scan

SECONDARY OUTCOMES:
Change in Positive and Negative Syndrome Scale | one hour after infusion to baseline
  Minimum: 30, Maximum: 210; higher score indicates worse outcome
Change in Brief Psychiatric Rating Scale | one hour after infusion to baseline
  Minimum: 18, Maximum: 126; higher score indicates worse outcome
Change in Clinician Administered Dissociative States Scale | one hour after infusion to baseline
  Minimum: 0, Maximum: 92; higher score indicates worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No